CLINICAL TRIAL: NCT06997614
Title: Enhancing Critical Thinking Competency and Nursing Quality in Critically Ill Patient Care: A Quasi-Experimental Study of an Evidence-Based Nutritional Management Protocol
Brief Title: Enhancing Critical Thinking Competency and Nursing Quality in Critically Ill Patient Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taizhou Hospital (Other)
Responsible Party: Principal Investigator, Yuexiang Zhao, Principal Investigator, Taizhou Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: No. 20240625
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2023-05

CONDITIONS: Evidence-Based Nursing; Critically Ill Patient; Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional group (Other): The conventional group adhered to conventional nutritional management methods and training
  Interventions: Other: Conventional group
- Evidence-based nursing group (Other): The study group implemented the EBN-based protocol alongside structured training
  Interventions: Other: evidence-based nursing group

INTERVENTIONS:
Other: Conventional group — The conventional group adhered to conventional nutritional management methods and training
  Arms: Conventional group
Other: evidence-based nursing group — The study group implemented the EBN-based protocol alongside structured training
  Arms: Evidence-based nursing group

SUMMARY:
The EBN-based nutritional management protocol effectively enhances junior nurses' specialized critical thinking competency and improves patient nutritional outcomes and satisfaction, demonstrating its potential to optimize critical care quality. However, further validation through multicenter studies with larger cohorts, extended follow-up periods, and additional outcome measures is warranted.

DETAILED DESCRIPTION:
This study aims to develop an evidence-based nursing (EBN)-based nutritional management protocol for critically ill patients and assess its effects on junior nurses' specialized critical thinking competency and nursing quality. A quasi-experimental design was employed, involving 7 junior nurses and 84 critically ill patients in each of the study and control groups. The study group implemented the EBN-based protocol alongside structured training, while the control group adhered to conventional practices. Nursing quality outcomes included assessments of nurses' specialized critical thinking skills, patient nutritional biomarkers (serum albumin, prealbumin), complication rates (aspiration, diarrhea, abdominal distension), and patient satisfaction. Multivariate binary logistic regression analysis identified influencing factors.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of critical illness by attending physicians or higher-qualified specialists according to established critical care diagnostic standards
* requirement for ICU admission with full access to standardized critical care and medical resources
* preserved partial gastrointestinal function without severe intestinal obstruction or perforation confirmed by certified nutritionists or senior nurses, enabling potential enteral nutrition (EN) or combined EN-parenteral nutrition (PN) support.

Exclusion Criteria:

* patients with severe cognitive impairment or psychiatric instability (e.g., advanced dementia, schizophrenia, status epilepticus) impairing capacity to engage in nutritional assessments or adhere to clinical protocols, which would jeopardize data collection reliability
* terminal-stage conditions (malignancies, renal/hepatic failure) with life expectancy < 7 days or exclusively receiving palliative care, leading to misalignment between their palliative nutritional goals and the study's therapeutic intervention objectives
* congenital metabolic disorders (e.g., phenylketonuria) or short bowel syndrome requiring specialized nutritional protocols, which were incompatible with conventional critical care nutritional protocols and could compromise the generalizability of study findings
* pregnancy/lactation due to unique nutritional demands and potential risks to fetal/infant development inherent in the study design, contravening established ethical standards
* cases involving transfer, voluntary discharge, or withdrawal of consent that compromised data completeness.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2022-11-05 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Improvement in Junior Nurses' Specialized Critical Thinking Competency | Baseline: Before training (Day 0). Post-intervention: 3 months after protocol implementation.
  Change in critical thinking scores measured by the Chinese Critical Thinking Disposition Inventory (CTDI-CV), a 70-item scale evaluating 7 dimensions (truth-seeking, open-mindedness, analyticity, systematicity, self-confidence, inquisitiveness, cognitive maturity) on a 6-point Likert scale. Higher scores indicate superior competency.

SECONDARY OUTCOMES:
Serum Albumin Levels | ICU admission (Day 0) and Day 14.
  Objective nutritional biomarker (g/L) measured via venous blood sampling.
Serum Prealbumin Levels | Day 0 and Day 14.
  Short-term nutritional status marker (mg/L) assessed alongside albumin.
Patient Satisfaction | Day 15.
  Self-reported satisfaction rated on a 5-point Likert scale (1: extremely dissatisfied, 5: extremely satisfied).

OTHER OUTCOMES:
Incidence of Aspiration | Daily monitoring until Day 14
  Binary outcome (yes/no) recorded during EN/PN administration.
Incidence of Diarrhea | Daily monitoring until Day 14.
  Defined as ≥3 loose stools/day, documented by nurses.
Incidence of Abdominal Distension | Daily monitoring until Day 14.
  Assessed via physical examination and patient reporting.
Body Weight Changes | Day 0 and Day 14.
  Measured in kg (bedside scales for ambulatory patients; estimated for others).
Blood Glucose Fluctuations Description: Time Frame: | Daily until Day 14
  Capillary/venous glucose levels (mmol/L) monitored per ICU protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- Taizhou Hospital of Traditional Chinese Medicine, Taizhou, Jiangsu, China